CLINICAL TRIAL: NCT03038035
Title: The Alzheimer's Disease THErapy With NEuroaid (ATHENE) Study : Assessing the Safety and Efficacy of Neuroaid II (MLC901) in Patients With Mild to Moderate Alzheimer's Disease Stable on Cholinesterase Inhibitors or Memantine: A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: The Alzheimer's Disease THErapy With NEuroaid (ATHENE) Study
Acronym: ATHENE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLC901-2
Record Dates: First submitted 2016-11-01; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuroaid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MLC901 (Active Comparator): NeuroAid II MLC901 is a derivative product of NeuroAid MLC601. It is a simplified formula based on the 9 Herbal ingredients that are present in NeuroAid MLC 601. Neuroaid II has been approved for sale as a Chinese Proprietary Medicine in Singapore by the HSA since March 2010. 24 weeks intervention. Dosage: 2 capsules 3 times a a day
  Upon completion of 24 weeks, subject will be given an option to continue an open-label extension for another 24 weeks.
  Interventions: Drug: MLC901
- Placebo (Placebo Comparator): 24 weeks intervention with orally placebo. 2 capsules 3 times a day.
  Upon completion of 24 weeks, subject will be given an option to continue an open-label extension for another 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MLC901 — 24 weeks intervention with orally MLC901. 2 capsules 3 times a day
  Other Names: Neuroaid II (MLC901)
  Arms: MLC901
Drug: Placebo — 24 weeks intervention with orally placebo. 2 capsules 3 times a day
  Other Names: MLC901 matched Placebo
  Arms: Placebo

SUMMARY:
MLC601 (Neuroaid) is a Traditional Chinese Medicine (TCM) having neuroprotective and neuroproliferative properties in cellular and animal models of brain injury. It contains 9 herbal and 5 non-herbal components. MLC901 (Neuroaid II), a simplified formula of MLC601, containing only the 9 herbal components yet showing the same efficacy has become available.

This study is carried out to find out if NEUROAID II (MLC901) is safe to be taken together with other established medicines for Alzheimer's disease and whether NEUROAID II (MLC901) helps in slowing down the Alzheimer's disease progression.

This study will be a 6-month randomized, double-blind, placebo-controlled trial, followed by an open extension study in which all subjects who completed the main 6 month trial (irrespective of treatment allocation) will be offered open-labelled MLC901 for another 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥50 years
* Diagnosed with probable AD according to NINCDS-ADRDA criteria,
* MMSE score of 10 to 24,
* Receiving the same AChEI or Memantine for the past 6 months prior to screening and on a stable dose for the past 4 months (stable dose is defined as 5 to 10mg/day for Donepezil, 3, 4.5 or 6 mg twice daily for rivastigmine capsules, 4.6 or 9.5 mg for rivastigmine transdermal patch once daily, 8 or 12 mg twice daily for galantamine tablets, 16 to 24 mg once daily for galantamine capsules XL, 10 mg OD or 10 mg BD for Memantine)
* Patient or legal representative is able to provide informed consent

Exclusion Criteria:

* Patients receiving any investigational product within 60 days or 5 half-lives prior to screening
* Any serious medical or psychiatric condition which in the investigator's judgement may jeopardize the patient by his/her participation in this study or may hamper his/her ability to perform and complete procedures required in the study.

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Evaluating the safety of MLC901 when it is given in combination with the standard treatment.The safety will be evaluated by adverse events, vital signs, ECG and laboratory tests, physical and neurological examinations at 6 months. | week 24

SECONDARY OUTCOMES:
Evaluate the effect of MLC901 as add on therapy to standard treatments for 6 months on cognitive function in patients with mild to moderate AD using Alzheimer's Disease Assessment Scale- cognitive subscale (ADAS- Cog). | week 24
Evaluate the effect of MLC901 as add on therapy to standard treatments for 6 months on cognitive function in patients with mild to moderate AD using Mini Mental State Examination (MMSE). | week 24
Evaluate the long term safety of MLC901 as add-on treatment to standard treatments for up to 1 year in an open extension study with adverse events, vital signs, ECG and laboratory tests, physical and neurological examination at 1 year. | week 48
Evaluate the long term effect on disease progression of MLC901 as add-on treatment to standard treatments for up to 1 year in an open extension study by assessing Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change (ADCS- CGIC). | week 48
  Using all of the other results (ADCS- ADL23, NPI, ADAS-Cog and MMSE) together would provide an accurate assessment of the disease progression.
Evaluate the long term effect on disease progression of MLC901 as add-on treatment to standard treatments for up to 1 year in an open extension study by assessing Alzheimer's Disease Cooperative Study- Activities of Daily Living Inventory (ADCS- ADL23) | week 48
  Using all of the other results (ADCS-CGIC, NPI, ADAS-Cog and MMSE) together would provide an accurate assessment of the disease progression.
Evaluate the long term effect on disease progression of MLC901 as add-on treatment to standard treatments for up to 1 year in an open extension study by assessing Neuropsychiatric Inventory (NPI). | week 48
  Using all of the other results (ADCS-CGIC, ADCS-ADL23, ADAS-Cog and MMSE) together would provide an accurate assessment of the disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Chen CLH, Lu Q, Moorakonda RB, Kandiah N, Tan BY, Villaraza SG, Cano J, Venketasubramanian N. Alzheimer's Disease THErapy With NEuroaid (ATHENE): A Randomized Double-Blind Delayed-Start Trial. J Am Med Dir Assoc. 2022 Mar;23(3):379-386.e3. doi: 10.1016/j.jamda.2021.10.018. Epub 2021 Nov 29. PMID 34856171